CLINICAL TRIAL: NCT05912127
Title: All On-4 Versus All o-3 Implant Treatment Concepts for Rehabilitation of Atrophied Mandibular Ridge. A Study of Patient Satisfaction
Brief Title: All on Four Versus All on Three Implant Treatment Concepts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A09071221
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Patients will be classified into 2 groups according to the implant treatment concept they received:
  * Group 1 (control group); included 3 patients who received All on 4 implant-supported fixed restoration. The patients received 2 inclined implants anterior to the mental foramina and 2 vertical implants in the lateral incisor/canine areas.
  * Group 2 (test group); included 3 patients who received All on 3 implant-supported fixed restoration. The patients received 2 inclined implants anterior to the mental foramina and 1 vertical implant in the midline of the mandible.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Group 1 (control group) (Active Comparator): patients who received All on 4 implant-supported fixed restoration. The patients received 2 inclined implants anterior to the mental foramina and 2 vertical implants in the lateral incisor/canine areas.
  Interventions: Device: implant supported fixed full arch prosthesis
- • Group 2 (test group); (Active Comparator): patients who received All on 3 implant-supported fixed restoration. The patients received 2 inclined implants anterior to the mental foramina and 1 vertical implant in the midline of the mandible.
  Interventions: Device: implant supported fixed full arch prosthesis

INTERVENTIONS:
Device: implant supported fixed full arch prosthesis — the patients will receive screw-retained cast metal-ceramic fixed prostheses that replace lost gingival tissues with pink porcelain.

SUMMARY:
the evaluation of patient satisfaction of All on-4 versus All on-3 implant treatment concepts rehabilitation of atrophied mandibular ridge.

DETAILED DESCRIPTION:
Patients will be classified into 2 groups according to the implant treatment concept they received:

* Group 1 (control group); included patients who received All on 4 implant-supported fixed restoration. The patients received 2 inclined implants anterior to the mental foramina and 2 vertical implants in the lateral incisor/canine areas.
* Group 2 (test group); included patients who received All on 3 implant-supported fixed restoration. The patients received 2 inclined implants anterior to the mental foramina and 1 vertical implant in the midline of the mandible.

ELIGIBILITY:
Inclusion Criteria:

* 1. All patients already have implants inserted in their mandibular ridges According to the All on 4 or All on 3 concepts.

  2. They were healthy, free from any systemic diseases relating to bone resorption such as uncontrolled diabetes or osteoporosis. This was achieved through medical history and clinical examination by the physician.

  3. All patients have sufficient inter-arch space. 4. All patients are of angle class I maxillo-mandibular relationships. 5. All patients had maxillary conventional complete dentures.

Exclusion Criteria:

1. Any neuromuscular disorders 2. Uncooperative patients

-

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-16 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2023-06-11 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | one year
  Patient satisfaction was evaluated using a questionnaire based on visual analog scale (VAS)
crestal bone loss | Two year
  bone loss was measured around the implants in mm

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Elsyad, professor, Principal Investigator — professor of prosthodontics, Faculty of dentistry , Mansoura University
Locations (1):
- Christine Ibrahim, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided